CLINICAL TRIAL: NCT01663467
Title: Efficacy of Internet and Smartphone Application-delivered TRT
Brief Title: Efficacy of Internet and Smartphone Application-delivered Tinnitus Retraining Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: there was no participants who were enrolled in this study
Sponsor: Seoul National University Hospital (Other)
Collaborators: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, YOUNG HO KIM, Associate Professor, Department of Otolaryngology-Head and Neck Surgery, Seoul National University College of Medicine, Seoul National University Boramae Medical Center, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUH_YHK_TRT
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Tinnitus
Keywords: tinnitus; smartphone; Web
MeSH Terms: conditions — Tinnitus | interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginkgo biloba only (Active Comparator): control group Ginexin-F 80mg tablet will be given twice a day for 6 months.
  Interventions: Drug: Ginkgo biloba
- Ginkgo biloba + modified TRT (Experimental): experimental group modified TRT (tinnitus retraining therapy) using smartphone and web based materials will be added with Ginkgo biloba.
  Ginexin-F 80mg tablet will be given twice a day for 6 months.
  Interventions: Drug: Ginkgo biloba; Behavioral: modified TRT

INTERVENTIONS:
Drug: Ginkgo biloba — Ginexin-F 80mg tablet will be given twice a day for 6 months.
  Other Names: Ginexin-F
Behavioral: modified TRT — modified TRT (tinnitus retraining therapy) using smartphone and web based materials will be added with Ginkgo biloba.
  Ginexin-F 80mg tablet will be given twice a day for 6 months.
  Arms: Ginkgo biloba + modified TRT

SUMMARY:
The purpose of this study is to prove the efficacy of the internet and smartphone application-delivered tinnitus retraining therapy (TRT).

DETAILED DESCRIPTION:
to investigate the effect of TRT with minimized counseling

ELIGIBILITY:
Inclusion Criteria:

* chronic subjective tinnitus

Exclusion Criteria:

* THI < 18

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 6 months
  THI will be evaluated 6 months after TRT using smatrphone and web

CONTACTS AND LOCATIONS:
Overall Officials: YOUNG HO KIM, MD., PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No